CLINICAL TRIAL: NCT01571284
Title: A Multicenter, Single Arm, Open Label Clinical Trial to Evaluate the Safety and Health-Related Quality of Life of Aflibercept in Patients With Metastatic Colorectal Cancer (mCRC) Previously Treated With an Oxaliplatin-Containing Regimen
Brief Title: Safety and Quality of Life Study of Aflibercept in Patients With Metastatic Colorectal Cancer Previously Treated With an Oxaliplatin-Based Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFLIBC06097; 2011-005724-17; U1111-1125-8949 (Other: UTN)
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — aflibercept; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin) (Experimental): Aflibercept 4 mg/kg IV infusion over 60 minutes followed by Irinotecan 180 mg/m^2 IV infusion over 90 minutes and Leucovorin 400 mg/m^2 IV infusion over 120 minutes at the same time followed by 5-Fluorouracil (5-FU) 400 mg/m^2 IV bolus over 2-4 minutes followed by 5-FU 2400 mg/m^2 continuous IV infusion over 46 hours on Day 1 of each cycle (1 Cycle = 2 weeks), until disease progression (DP), unacceptable toxicity, death, Investigator's decision or participant's refusal of further treatment.
  Interventions: Drug: AFLIBERCEPT AVE0005; Drug: FOLFIRI

INTERVENTIONS:
Drug: AFLIBERCEPT AVE0005 — Pharmaceutical form:Concentrate for solution for infusion Route of administration: Intravenous
Drug: FOLFIRI — irinotecan, 5-FU and leucovorin

SUMMARY:
Primary Objective:

To provide metastatic colorectal cancer participants with access to aflibercept and to document the overall safety in these participants

Secondary Objective:

To document the Health-Related Quality of Life of aflibercept in this participants population

DETAILED DESCRIPTION:
Each participants will be treated until disease progression, unacceptable toxicity, death, Investigator's decision or participant's refusal for further treatment (whichever comes first). Participants were followed-up during study treatment and for at least 30 days after last administration.

ELIGIBILITY:
Inclusion criteria :

* Histologically or cytologically proven adenocarcinoma of the colon or rectum.
* Metastatic disease.
* Eastern Cooperative Oncology Group performance status 0-1.
* One and only one prior chemotherapeutic regimen for metastatic disease. This prior chemotherapy was an oxaliplatin containing regimen. Participants must had progressed during or after the oxaliplatin based chemotherapy. Participants relapsed within 6 months of completion of oxaliplatin adjuvant chemotherapy were eligible.
* Signed written informed consent obtained prior to inclusion.

Exclusion criteria:

* Prior therapy with irinotecan.
* Inadequate bone marrow, liver and renal function: neutrophils < 1.5x109/L, platelets < 100x109/L, hemoglobin < 9.0 g/dL, total bilirubin >1.5 x upper normal limit (ULN), transaminases >3 x ULN (unless liver metastasis are present), alkaline phosphatase >3 x ULN (unless liver metastasis are present), serum creatinine > 1.5 x ULN.
* Less than 4 weeks from prior radiotherapy, prior chemotherapy, prior major surgery (or until the surgical wound were fully healed).
* Treatment with any investigational drug within the prior 30 days.
* Treatment with concomitant anticonvulsivant agents that were CYP3A4 inducers (phenytoin, phenobarbital, carbamazepine), unless discontinued >7 days.
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease.
* Prior malignancy (other than colorectal) including prior malignancy from which the participants had been disease free for < 5 years (except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix).
* Any of the following within 6 months prior to study inclusion: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, severe congestive heart failure, stroke or transient ischemic attack.
* Any of the following within 3 months prior study inclusion: severe gastrointestinal bleeding/hemorrhage, treatment resistant peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event.
* Occurrence of deep vein thrombosis within 4 weeks, prior to study inclusion.
* Known acquired immunodeficiency syndrome (AIDS-related illnesses) or known HIV disease requiring antiretroviral treatment.
* Known dihydropyrimidine dehydrogenase deficiency.
* Predisposing colonic or small bowel disorders in which the symptoms were uncontrolled.
* Prior history of chronic enteropathy, inflammatory enteropathy, chronic diarrhea, unresolved bowel obstruction/sub-obstruction, more than hemicolectomy, extensive small intestine resection with chronic diarrhea.
* Known Gilbert's syndrome.
* Unresolved or unstable toxicity from any prior anti cancer therapy at the time of inclusion.
* History of anaphylaxis or known intolerance to atropine sulphate or loperamide or appropriate antiemetics to be administered in conjunction with FOLFIRI (irinotecan, 5-Fluorouracil, leucovorin).
* Severe acute or chronic medical condition, which could impair the ability of the participants to participate to the study.
* Urine protein-creatinine ratio (UPCR) >1 on morning spot urinalysis or proteinuria > 500 mg/24-h.
* Uncontrolled hypertension within 3 months prior to study inclusion.
* Participants on anticoagulant therapy with unstable dose of warfarin and/or had an out-of-therapeutic range INR within the 4 weeks prior to study inclusion.
* Evidence of clinically significant bleeding predisposition or underlying coagulopathy, non-healing wound.
* Pregnant or breast-feeding women.
* Participants with reproductive potential who were not agree to use an accepted effective method of contraception.

The above information wass not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2012-05-30 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (179):
- United States (12):
  - Investigational Site Number 840-002, Muscle Shoals, Alabama
  - Investigational Site Number 840-008, Corona, California
  - Investigational Site Number 840-007, Fountain Valley, California
  - Investigational Site Number 840-004, Riverside, California
  - Investigational Site Number 840-006, Indianapolis, Indiana
  - Investigational Site Number 840-011, Metairie, Louisiana
  - Investigational Site Number 840-001, Rockville, Maryland
  - Investigational Site Number 840-010, Howell Township, New Jersey
  - Investigational Site Number 840-012, Albuquerque, New Mexico
  - Investigational Site Number 840-009, Farmington, New Mexico
  - Investigational Site Number 840-003, Lake Success, New York
  - Investigational Site Number 840-005, Middletown, Ohio
- Belgium (12):
  - Investigational Site Number 056010, Aalst
  - Investigational Site Number 056015, Arlon
  - Investigational Site Number 056004, Bonheiden
  - Investigational Site Number 056001, Edegem
  - Investigational Site Number 056012, Ghent
  - Investigational Site Number 056009, Haine-Saint-Paul
  - Investigational Site Number 056003, Liège
  - Investigational Site Number 056007, Liège
  - Investigational Site Number 056014, Loverval
  - Investigational Site Number 056013, Turnhout
  - Investigational Site Number 056002, Verviers
  - Investigational Site Number 056011, Yvoir
- Brazil (11):
  - Investigational Site Number 008, Brasília
  - Investigational Site Number 009, Curitiba
  - Investigational Site Number 012, Fortaleza
  - Investigational Site Number 006, Passo Fundo
  - Investigational Site Number 003, Porto Alegre
  - Investigational Site Number 002, Rio de Janeiro
  - Investigational Site Number 011, Salvador
  - Investigational Site Number 013, São José do Rio Preto
  - Investigational Site Number 001, São Paulo
  - Investigational Site Number 004, São Paulo
  - Investigational Site Number 005, São Paulo
- Canada (6):
  - Investigational Site Number 124002, Calgary
  - Investigational Site Number 124003, Montreal
  - Investigational Site Number 124005, Montreal
  - Investigational Site Number 124004, Ottawa
  - Investigational Site Number 124006, Québec
  - Investigational Site Number 124001, Toronto
- Chile (2):
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152003, Santiago
- Czechia (6):
  - Investigational Site Number 203005, Brno
  - Investigational Site Number 203003, Olomouc
  - Investigational Site Number 203001, Ostrava
  - Investigational Site Number 203002, Prague
  - Investigational Site Number 203004, Prague
  - Investigational Site Number 203006, Zlín
- Denmark (3):
  - Investigational Site Number 208001, Cph Ø
  - Investigational Site Number 208003, Hillerød
  - Investigational Site Number 208002, Odense C
- Finland (2):
  - Investigational Site Number 246001, Oulu
  - Investigational Site Number 246002, Turku
- Germany (20):
  - Investigational Site Number 276-016, Aschaffenburg
  - Investigational Site Number 276-010, Augsburg
  - Investigational Site Number 276-011, Berlin
  - Investigational Site Number 276-012, Erlangen
  - Investigational Site Number 276-009, Frankfurt am Main
  - Investigational Site Number 276-013, Frankfurt am Main
  - Investigational Site Number 276-004, Halle
  - Investigational Site Number 276-007, Krefeld
  - Investigational Site Number 276-003, Lebach
  - Investigational Site Number 276-019, Leipzig
  - Investigational Site Number 276-008, Ludwigsburg
  - Investigational Site Number 276-018, Magdeburg
  - Investigational Site Number 276-014, Magdeburg
  - Investigational Site Number 276-006, Moers
  - Investigational Site Number 276-001, München
  - Investigational Site Number 276-002, München
  - Investigational Site Number 276-015, Northeim
  - Investigational Site Number 276-017, Velbert
  - Investigational Site Number 276-005, Weiden/Oberpfalz
  - Investigational Site Number 276-020, Wolfsburg
- Ireland (3):
  - Investigational Site Number 372002, Dublin
  - Investigational Site Number 372004, Galway
  - Investigational Site Number 372001, Wilton
- Israel (5):
  - Investigational Site Number 376002, Haifa
  - Investigational Site Number 376001, Jerusalem
  - Investigational Site Number 376005, Petah Tikva
  - Investigational Site Number 376003, Tel Aviv
  - Investigational Site Number 376004, Tel Litwinsky
- Italy (28):
  - Investigational Site Number 380-005, Ancona
  - Investigational Site Number 380-029, Bergamo
  - Investigational Site Number 380-021, Bologna
  - Investigational Site Number 380-004, Brescia
  - Investigational Site Number 380-007, Candiolo
  - Investigational Site Number 380-012, Catania
  - Investigational Site Number 380-019, Catanzaro
  - Investigational Site Number 380-023, Florence
  - Investigational Site Number 380-001, Genova
  - Investigational Site Number 380-014, Meldola
  - Investigational Site Number 380-016, Messina
  - Investigational Site Number 380-013, Milan
  - Investigational Site Number 380-015, Milan
  - Investigational Site Number 380-025, Milan
  - Investigational Site Number 380-022, Napoli
  - Investigational Site Number 380-028, Novara
  - Investigational Site Number 380-017, Padua
  - Investigational Site Number 380-002, Pisa
  - Investigational Site Number 380-008, Reggio Emilia
  - Investigational Site Number 380-024, Roma
  - Investigational Site Number 380-010, Roma
  - Investigational Site Number 380-011, Roma
  - Investigational Site Number 380-006, San Giovanni Rotondo
  - Investigational Site Number 380-026, Sassari
  - Investigational Site Number 380-020, Terni
  - Investigational Site Number 380-009, Torino
  - Investigational Site Number 380-003, Udine
  - Investigational Site Number 380-018, Verona
- Investigational Site Number 1, Beirut, Lebanon
- Mexico (4):
  - Investigational Site Number 484002, Mexico City
  - Investigational Site Number 484009, Mexico City
  - Investigational Site Number 484010, México, D.F.
  - Investigational Site Number 484001, Monterrey
- Netherlands (2):
  - Investigational Site Number 528001, Hoofddorp
  - Investigational Site Number 528002, Zwolle
- Norway (2):
  - Investigational Site Number 578002, Bergen
  - Investigational Site Number 578001, Oslo
- Investigational Site Number 630-001, Rio Peidras, Puerto Rico
- Russia (7):
  - Investigational Site Number 643003, Kazan'
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643004, Moscow
  - Investigational Site Number 643005, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643006, Moscow
  - Investigational Site Number 643009, Saint Petersburg
- Spain (16):
  - Investigational Site Number 724016, Alicante
  - Investigational Site Number 724008, Barakaldo
  - Investigational Site Number 724012, Cáceres
  - Investigational Site Number 724002, Córdoba
  - Investigational Site Number 724013, Donostia / San Sebastian
  - Investigational Site Number 724014, L'Hospitalet de Llobregat
  - Investigational Site Number 724003, Madrid
  - Investigational Site Number 724015, Madrid
  - Investigational Site Number 724005, Madrid
  - Investigational Site Number 724004, Málaga
  - Investigational Site Number 724010, Sabadell
  - Investigational Site Number 724011, Santander
  - Investigational Site Number 724006, Santiago de Compostela
  - Investigational Site Number 724001, Valencia
  - Investigational Site Number 724009, Valencia
  - Investigational Site Number 724007, Zaragoza
- Sweden (2):
  - Investigational Site Number 752_002, Jönköping
  - Investigational Site Number 752_001, Vaxjo
- Thailand (10):
  - Investigational Site Number 764002, Bangkok
  - Investigational Site Number 764003, Bangkok
  - Investigational Site Number 764008, Bangkok
  - Investigational Site Number 764001, Bangkok
  - Investigational Site Number 764006, Bangkok
  - Investigational Site Number 764005, Bangkok,TH
  - Investigational Site Number 764009, Chiang Mai
  - Investigational Site Number 764004, Khon Kaen
  - Investigational Site Number 764010, Laksi
  - Investigational Site Number 764007, Lopburi
- Turkey (Türkiye) (12):
  - Investigational Site Number 792-06, Adana
  - Investigational Site Number 792-01, Ankara
  - Investigational Site Number 792-09, Ankara
  - Investigational Site Number 792-08, Ankara
  - Investigational Site Number 792-02, Çapa
  - Investigational Site Number 792010, Edirne
  - Investigational Site Number 792-05, Gaziantep
  - Investigational Site Number 792012, Istanbul
  - Investigational Site Number 792-03, Istanbul
  - Investigational Site Number 792-04, Istanbul
  - Investigational Site Number 792-007, Izmir
  - Investigational Site Number 792011, Izmir
- United Kingdom (12):
  - Investigational Site Number 826005, Dudley
  - Investigational Site Number 826011, Hull
  - Investigational Site Number 826008, Leicester
  - Investigational Site Number 826007, London
  - Investigational Site Number 826012, London
  - Investigational Site Number 826003, Maidstone
  - Investigational Site Number 826009, Manchester
  - Investigational Site Number 826004, Newcastle upon Tyne
  - Investigational Site Number 826006, Northwood
  - Investigational Site Number 826002, Southampton
  - Investigational Site Number 826001, Sutton
  - Investigational Site Number 826010, Taunton

REFERENCES:
- [Derived] Riechelmann RP, Srimuninnimit V, Bordonaro R, Kavan P, Di Bartolomeo M, Maiello E, Cicin I, Garcia-Alfonso P, Chau I, Fedyanin MY, Martos CF, Ter-Ovanesov M, Peeters M, Ko YJ, Yalcin S, Karthaus M, Aparicio J, Heinemann V, Picard P, Bury D, Drea E, Sobrero A. Aflibercept Plus FOLFIRI for Second-line Treatment of Metastatic Colorectal Cancer: Observations from the Global Aflibercept Safety and Health-Related Quality-of-Life Program (ASQoP). Clin Colorectal Cancer. 2019 Sep;18(3):183-191.e3. doi: 10.1016/j.clcc.2019.05.003. Epub 2019 May 15. PMID 31221542

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 151 sites in 23 countries. A total of 798 participants were screened between 30 May 2012 and 03 January 2015, out of which 781 participants were enrolled and 779 participants were treated.
Pre-assignment Details: Participants enrolled in the study to assess the safety of Aflibercept in participants treated with a combination of Aflibercept with FOLFIRI regimen (Irinotecan, Leucovorin and 5-Fluorouracil [5-FU]).
Groups:
- Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin): Aflibercept 4 mg/kg intravenous (IV) infusion over 60 minutes followed by Irinotecan 180 mg/m^2 IV infusion over 90 minutes and Leucovorin 400 mg/m^2 IV infusion over 120 minutes at the same time followed by 5-FU 400 mg/m^2 IV bolus over 2-4 minutes followed by 5-FU 2400 mg/m^2 continuous IV infusion over 46 hours on Day 1 of each cycle (1 Cycle = 2 weeks), until disease progression (DP), unacceptable toxicity, death, Investigator's decision or participant's refusal of further treatment.
Period: Overall Study
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Started | 781
Safety Population (Participants who signed informed consent form and received at least part of one dose of treatment.) | 779
Completed | 612 (403 participants with DP and 209 with adverse events were considered as completed.)
Not Completed | 169
Not completed — Participant's decision | 84
Not completed — Lost to Follow-up | 3
Not completed — Enrolled but not treated | 2
Not completed — Other than specified above | 80

BASELINE CHARACTERISTICS:
Population: Safety population defined as the participants who signed the informed consent form and received at least part of one dose of study treatment.
Groups:
- Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin): Aflibercept 4 mg/kg IV infusion over 60 minutes followed by Irinotecan 180 mg/m^2 IV infusion over 90 minutes and Leucovorin 400 mg/m^2 IV infusion over 120 minutes at the same time followed by 5-FU 400 mg/m^2 IV bolus over 2-4 minutes followed by 5-FU 2400 mg/m^2 continuous IV infusion over 46 hours on Day 1 of each cycle (1 Cycle = 2 weeks), until DP, unacceptable toxicity, death, Investigator's decision or participant's refusal of further treatment.
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314
  Male | 465
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 631
  Black or African | 8
  American Asian | 121
  Other | 19
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.80 (0.23)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Number of participants analyzed = participants with available data for specified measure.
  mmHg
    number analyzed (Participants) | 776
    (all) | 126.4 (13.4)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Number of participants analyzed = participants with available data for specified measure.
  mmHg
    number analyzed (Participants) | 776
    (all) | 76.4 (9.0)
Any Relevant Medical/Surgical History [Count of Participants; unit: Participants] — Any relevant medical/surgical history including detailed cardiovascular risk factors and prior vascular events if any.
  Participants | 640
History of Thrombovascular Event and/or Presence of Cardiovascular Risk Factor [Count of Participants; unit: Participants] | 424
Time From Initial Histological Diagnosis till Baseline Visit [Mean (Standard Deviation); unit: Months] | 19.1 (17.2)
Location of Primary Tumor [Count of Participants; unit: Participants]
  Colon | 406
  Recto sigmoid | 171
  Rectum | 200
  Other | 2
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 778
  Other | 1
Organs with Metastases at Baseline [Count of Participants; unit: Participants]
  1 | 358
  >1 | 421
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS is used to assess how the disease affects the daily living abilities of the participant. It ranges on the scale from 0-5 (0= normal activity; 1= symptoms but ambulatory; 2= in bed for less than (<) 50 percent (%) of the time; 3= in bed for greater than (>) 50% of the time; 4= 100% bedridden; 5= dead.
  Participants
    0 | 484
    1 | 292
    Missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an adverse event (AE) without regard to possibility of causal relationship with this treatment. A serious AE (SAE): Any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs. National Cancer Institute Common Terminology Criteria (NCI-CTCAE) Version 4.03 was used to assess severity (Grade 1=mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening/disabling) of AEs.
Time Frame: Baseline up to 30 days after the last treatment administration (either Aflibercept or FOLFIRI whichever comes last) (maximum exposure: 214 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  Any TEAE (All Grades) | 769
  Any TEAEs (Grades 3-4) | 609
  Any serious TEAE | 272
  Any serious related TEAE | 159
  Any TEAE leading to death | 47
  Any TEAE (permanent treatment discontinuation) | 208
  Any TEAE (premature treatment discontinuation) | 104

2. Primary Outcome: Number of Participants With Abnormal Hematological Parameters
Description: Abnormal hematological parameters included: anaemia, thrombocytopenia, leukopenia and neutropenia. Number of participants with each of these parameters were analyzed by grades (All Grades and Grades 3-4 as per NCI CTCAE (Version 4.03), where Grade 1=mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening/disabling. All Grades included Grades 1-4.
Time Frame: as for outcome 1
Population: Safety population. Here, 'Number Analyzed = participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  Anaemia: All Grades: number analyzed (Participants) | 744
  Anaemia: All Grades | 535
  Anaemia: Grades 3-4: number analyzed (Participants) | 744
  Anaemia: Grades 3-4 | 14
  Thrombocytopenia: All Grades: number analyzed (Participants) | 745
  Thrombocytopenia: All Grades | 293
  Thrombocytopenia: Grades 3-4: number analyzed (Participants) | 745
  Thrombocytopenia: Grades 3-4 | 13
  Leukopenia: All Grades: number analyzed (Participants) | 745
  Leukopenia: All Grades | 532
  Leukopenia: Grades 3-4: number analyzed (Participants) | 745
  Leukopenia: Grades 3-4 | 72
  Neutropenia: All Grades: number analyzed (Participants) | 744
  Neutropenia: All Grades | 450
  Neutropenia: Grades 3-4: number analyzed (Participants) | 744
  Neutropenia: Grades 3-4 | 227

3. Primary Outcome: Number of Participants With International Normalized Ratio (INR)
Description: The INR is a derived measure of the prothrombin time. The INR is the ratio of a participant's prothrombin time to a normal control sample. Normal range (without anti coagulation therapy): 0.8-1.2; Targeted range (with anti coagulation therapy) 2.0-3.0.
Time Frame: as for outcome 1
Population: Safety population. Here, 'Number Analyzed' = participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  INR<1.5: number analyzed (Participants) | 110
  INR<1.5 | 106
  INR>=1.5 to <3: number analyzed (Participants) | 110
  INR>=1.5 to <3 | 0
  INR>=3 to <5: number analyzed (Participants) | 110
  INR>=3 to <5 | 2
  INR>=5: number analyzed (Participants) | 110
  INR>=5 | 2

4. Primary Outcome: Number of Participants With Abnormal Electrolytes Parameters
Description: Abnormal electrolytes parameters included: hyponatremia, hypernatremia, hypocalcemia, hypercalcemia, hypokalemia, and hyperkalemia. Number of participants with each of these parameters were analyzed by grades ( All Grades and Grades 3-4 as per NCI CTCAE Version 4.03, where Grade 1=mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening/disabling. All Grades included Grades 1-4.
Time Frame: as for outcome 1
Population: Safety population. Here, 'Number Analyzed' = participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  Hyponatremia: All Grades: number analyzed (Participants) | 736
  Hyponatremia: All Grades | 181
  Hyponatremia: Grades 3-4: number analyzed (Participants) | 736
  Hyponatremia: Grades 3-4 | 32
  Hypernatremia: All Grades: number analyzed (Participants) | 736
  Hypernatremia: All Grades | 75
  Hypernatremia: Grades 3-4: number analyzed (Participants) | 736
  Hypernatremia: Grades 3-4 | 1
  Hypocalcemia: All Grades: number analyzed (Participants) | 682
  Hypocalcemia: All Grades | 213
  Hypocalcemia: Grades 3-4: number analyzed (Participants) | 682
  Hypocalcemia: Grades 3-4 | 5
  Hypercalcemia: All Grades: number analyzed (Participants) | 682
  Hypercalcemia: All Grades | 52
  Hypercalcemia: Grades 3-4: number analyzed (Participants) | 682
  Hypercalcemia: Grades 3-4 | 2
  Hypokalemia: All Grades: number analyzed (Participants) | 734
  Hypokalemia: All Grades | 121
  Hypokalemia: Grades 3-4: number analyzed (Participants) | 734
  Hypokalemia: Grades 3-4 | 16
  Hyperkalemia: All Grades: number analyzed (Participants) | 734
  Hyperkalemia: All Grades | 166
  Hyperkalemia: Grades 3-4: number analyzed (Participants) | 734
  Hyperkalemia: Grades 3-4 | 10

5. Primary Outcome: Number of Participants With Abnormal Renal and Liver Function Parameters
Description: Renal and liver function parameters included: creatinine, hyperbilirubinemia, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase. Number of participants with each of these parameters were analyzed by grades (All Grades and Grades 3-4) as per NCI CTCAE version 4.03, where Grade 1=mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening/disabling. All Grades included Grades 1-4.
Time Frame: as for outcome 1
Population: Safety population. Here, 'Number Analyzed' = participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  Creatinine: All Grades: number analyzed (Participants) | 737
  Creatinine: All Grades | 161
  Creatinine: Grades 3-4: number analyzed (Participants) | 737
  Creatinine: Grades 3-4 | 2
  Hyperbilirubinemia: All Grades: number analyzed (Participants) | 734
  Hyperbilirubinemia: All Grades | 130
  Hyperbilirubinemia: Grades 3-4: number analyzed (Participants) | 734
  Hyperbilirubinemia: Grades 3-4 | 9
  AST: All Grades: number analyzed (Participants) | 727
  AST: All Grades | 342
  AST: Grades 3-4: number analyzed (Participants) | 727
  AST: Grades 3-4 | 12
  ALT: All Grades: number analyzed (Participants) | 736
  ALT: All Grades | 270
  ALT: Grades 3-4: number analyzed (Participants) | 736
  ALT: Grades 3-4 | 10
  Alkaline phosphatase: All Grades: number analyzed (Participants) | 733
  Alkaline phosphatase: All Grades | 465
  Alkaline phosphatase: Grades 3-4: number analyzed (Participants) | 733
  Alkaline phosphatase: Grades 3-4 | 23

6. Primary Outcome: Creatinine Clearance of Aflibercept Plus FOLFIRI
Description: Creatinine clearance is a measure of kidney function. Creatinine clearance rate is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Creatinine clearance can be measured directly or estimated using established formulas. For this study, the creatinine clearance was calculated using the Cockroft-Gault or Modification of Diet in Renal Disease (MDRD).
Time Frame: as for outcome 1
Population: Safety population. Overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 312
mL/min | 71.4 (29.3)

7. Primary Outcome: Number of Participants With Other Abnormal Biochemistry Parameters
Description: Other abnormal biochemistry parameters included: hypoglycemia, hyperglycemia and hypoalbuminemia. Number of participants with each of these parameters were analyzed by grades (All Grades and Grades 3-4) as per NCI CTCAE Version 4.03, where Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening/disabling. All Grades included Grades 1-4.
Time Frame: as for outcome 1
Population: Safety population. Here, 'Number Analyzed' = participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  Hypoglycemia: All Grades: number analyzed (Participants) | 725
  Hypoglycemia: All Grades | 90
  Hypoglycemia: Grades 3-4: number analyzed (Participants) | 725
  Hypoglycemia: Grades 3-4 | 6
  Hyperglycemia: All Grades: number analyzed (Participants) | 725
  Hyperglycemia: All Grades | 403
  Hyperglycemia: Grades 3-4: number analyzed (Participants) | 725
  Hyperglycemia: Grades 3-4 | 30
  Hypoalbuminemia: All Grades: number analyzed (Participants) | 689
  Hypoalbuminemia: All Grades | 241
  Hypoalbuminemia: Grades 3-4: number analyzed (Participants) | 689
  Hypoalbuminemia: Grades 3-4 | 6

8. Primary Outcome: Number of Participants With Abnormal Non-Gradable Biochemistry Parameters
Description: Non-gradeable biochemistry parameters included; chloride, urea, total protein, blood urea nitrogen (BUN) and lactate dehydrogenase (LDH). Number of participants with <lower limit of normal ranges (LLN) and >upper limit of normal ranges (ULN) for each of these parameters were reported.
Time Frame: as for outcome 1
Population: Safety population. Here, 'Number Analyzed = participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  Chloride<LLN: number analyzed (Participants) | 711
  Chloride<LLN | 135
  Chloride>ULN: number analyzed (Participants) | 711
  Chloride>ULN | 217
  BUN<LLN: number analyzed (Participants) | 258
  BUN<LLN | 41
  BUN>ULN: number analyzed (Participants) | 258
  BUN>ULN | 83
  UREA<LLN: number analyzed (Participants) | 591
  UREA<LLN | 60
  UREA>ULN: number analyzed (Participants) | 591
  UREA>ULN | 250
  LDH<LLN: number analyzed (Participants) | 723
  LDH<LLN | 79
  LDH>ULN: number analyzed (Participants) | 723
  LDH>ULN | 423
  Total proteins<LLN: number analyzed (Participants) | 711
  Total proteins<LLN | 162
  Total proteins>ULN: number analyzed (Participants) | 711
  Total proteins>ULN | 77

9. Primary Outcome: Number of Participants With Proteinuria Events
Description: Proteinuria is defined as the ratio of protein to creatinine. Number of participants with proteinuria were analyzed by grades (Grades 1, 2, 3 ,4) as per NCI CTCAE Version 4.03 where Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening/disabling.
Time Frame: as for outcome 1
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  Grade 1 | 286
  Grade 2 | 123
  Grade 3 | 54
  Grade 4 | 5

10. Primary Outcome: Number of Participants With Proteinuria Grade >=2
Description: Proteinuria is defined as the ratio of protein to creatinine. Number of participants with proteinuria grade >=2 (graded as per NCI CTCAE Version 4.03), where Grade>=2 represents moderate to life-threatening/disabling event.
Time Frame: as for outcome 1
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
participants | 182

11. Primary Outcome: Number of Participants With Urinary Protein-Creatinine Ratio (UPCR)
Description: Urinary protein creatinine ratio (UPCR) corresponds to the ratio of the urinary protein and urinary creatinine concentration (expressed in mg/dL). This ratio provides an accurate quantification of 24-hours urinary protein excretion. There is a high correlation between morning UPCR and 24-hour proteinuria in participants with normal or reduced renal functions. Normal ratio is < or = 1.
Time Frame: as for outcome 1
Population: Safety population. Here, 'Number Analyzed = participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  UPCR<=1: number analyzed (Participants) | 367
  UPCR<=1 | 265
  UPCR>=1 to <=2: number analyzed (Participants) | 367
  UPCR>=1 to <=2 | 51
  UPCR>=2 to <=3: number analyzed (Participants) | 367
  UPCR>=2 to <=3 | 24
  UPCR>3: number analyzed (Participants) | 367
  UPCR>3 | 27

12. Primary Outcome: Number of Participants With Proteinuria (Grade>=2) Concomitant With Hematuria and /or Hypertension
Description: Proteinuria is defined as the presence of excess proteins in the urine (assessed either by spot sample, dipstick/ urine protein or 24 hour urine collection). Hematuria is defined as the presence of blood in urine (positive dipstick for RBC or reported AE). Number of participants with proteinuria grade >=2 (graded as per NCI CTCAE Version 4.03), where Grade>=2 represents moderate to life-threatening/disabling event. Hypertension (high blood pressure) is defined as having a blood pressure reading of more than 140/90 mmHg over a number of weeks.
Time Frame: as for outcome 1
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  Proteinuria with hematuria | 72
  Proteinuria with hypertension | 4
  Proteinuria with hematuria and hypertension | 3

13. Primary Outcome: Number of Participants With Cycle Delay and/or Dose Modification
Description: A theoretical cycle is a 2 week period i.e. 14 days. A cycle is delayed if duration of previous cycle is greater than 14+2 days ; dose modification includes dose reduction and dose omission.
Time Frame: as for outcome 1
Population: Safety population defined as the participants who signed the informed consent form and received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 779
Participants
  No delay and no dose modification | 119
  Any delay and/or dose modification | 660
  Delay only | 163
  Delay and Aflibercept modified | 39
  Delay and FOLFIRI modified | 308
  Delay and Aflibercept and Folfiri modified | 97
  Only Aflibercept modified | 5
  Only FOLFIRI modified | 43
  Both Aflibercept and FOLFIRI modified | 5

14. Secondary Outcome: Mean Change From Baseline in Health Related Quality of Life (HRQL) European Organization for Research and Treatment for Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30 Score): Global Health Status
Description: EORTC-QLQ-C30 is a cancer-specific instrument with 30 questions for evaluation of new chemotherapy and provides an assessment of participant reported outcome dimensions. First 28 questions used 4-point scale (1=not at all,2=a little,3=quite a bit,4=very much) for evaluating 5 functional scales (physical,role,emotional,cognitive,social), 3 symptom scales (fatigue,nausea/vomiting,pain) & other single items. For each item,high score represented high level of symptomatology/problem. Last 2 questions represented participant's assessment of overall health & quality of life, coded on 7-point scale (1=very poor to 7=excellent).EORTC QLQ-C30 observed values and change from baseline for global health status (scoring of questions 29 & 30) and 5 functional scales, 3 symptom scales and other single items (scoring of questions 1 to 28). Answers were converted into grading scale, with values between 0 and 100. A high score represented a favourable outcome with a best quality of life for participant.
Time Frame: Pre-dose at Baseline, Day 1 of every odd cycle (from Cycle 3 to 35); at the end of treatment (EOT) (within 30 days of last treatment) (maximum exposure: 214 weeks)
Population: EORTC QLQ-C30 analysis population: participants who signed informed consent form; had an evaluable QLQ-C30 questionnaire at baseline and at least one evaluable assessment post baseline and received at least part of one dose of study treatment (either Aflibercept or FOLFIRI). Here, 'Number Analyzed' = participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 636
units on a scale
  Baseline: number analyzed (Participants) | 630
  Baseline | 68.61 (20.48)
  Change at Cycle 3: number analyzed (Participants) | 549
  Change at Cycle 3 | -3.34 (18.83)
  Change at Cycle 5: number analyzed (Participants) | 429
  Change at Cycle 5 | -4.70 (18.89)
  Change at Cycle 7: number analyzed (Participants) | 344
  Change at Cycle 7 | -3.63 (22.02)
  Change at Cycle 9: number analyzed (Participants) | 273
  Change at Cycle 9 | -3.97 (21.31)
  Change at Cycle 11: number analyzed (Participants) | 232
  Change at Cycle 11 | -5.85 (22.26)
  Change at Cycle 13: number analyzed (Participants) | 151
  Change at Cycle 13 | -2.26 (21.69)
  Change at Cycle 15: number analyzed (Participants) | 123
  Change at Cycle 15 | -3.05 (22.46)
  Change at Cycle 17: number analyzed (Participants) | 85
  Change at Cycle 17 | -1.18 (22.50)
  Change at Cycle 19: number analyzed (Participants) | 60
  Change at Cycle 19 | -2.36 (22.92)
  Change at Cycle 21: number analyzed (Participants) | 45
  Change at Cycle 21 | -5.56 (23.77)
  Change at Cycle 23: number analyzed (Participants) | 34
  Change at Cycle 23 | -6.86 (19.94)
  Change at Cycle 25: number analyzed (Participants) | 29
  Change at Cycle 25 | -8.05 (16.89)
  Change at Cycle 27: number analyzed (Participants) | 23
  Change at Cycle 27 | -10.14 (17.58)
  Change at Cycle 29: number analyzed (Participants) | 20
  Change at Cycle 29 | -8.33 (14.05)
  Change at Cycle 31: number analyzed (Participants) | 15
  Change at Cycle 31 | -9.44 (16.92)
  Change at Cycle 33: number analyzed (Participants) | 11
  Change at Cycle 33 | -11.36 (21.82)
  Change at Cycle 35: number analyzed (Participants) | 10
  Change at Cycle 35 | -5.83 (20.81)
  Change at EOT: number analyzed (Participants) | 340
  Change at EOT | -8.82 (23.95)

15. Secondary Outcome: Mean Change From Baseline in HRQL EORTC QLQ-C30 Score: Functional Scales
Description: EORTC-QLQ-C30 is a cancer-specific instrument with 30 questions for evaluation of new chemotherapy and provides an assessment of participant reported outcome dimensions. First 28 questions used 4-point scale (1=not at all,2=a little,3=quite a bit,4=very much) for evaluating 5 functional scales (physical,role,emotional,cognitive,social), 3 symptom scales (fatigue,nausea/vomiting,pain) & other single items. For each item,high score represented high level of symptomatology/problem. Last 2 questions represented participant's assessment of overall health & quality of life, coded on 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 observed values and change from baseline for global health status (scoring of questions 29 & 30) and 5 functional scales, 3 symptom scales and other single items (scoring of questions 1 to 28).Answers were converted into grading scale, with values between 0 and 100. A high score represented a favourable outcome with a best quality of life for participant.
Time Frame: Pre-dose at Baseline, Day 1 of every odd cycle (from Cycle 3 to 35); at EOT (within 30 days of last treatment) (maximum exposure: 214 weeks)
Population: EORTC QLQ-C30 analysis population. Here, 'Number Analyzed' = participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 636
units on a scale
  Physical - Baseline: number analyzed (Participants) | 634
  Physical - Baseline | 81.79 (19.41)
  Physical - Change at Cycle 3: number analyzed (Participants) | 551
  Physical - Change at Cycle 3 | -3.73 (15.15)
  Physical - Change at Cycle 5: number analyzed (Participants) | 439
  Physical - Change at Cycle 5 | -3.95 (15.22)
  Physical - Change at Cycle 7: number analyzed (Participants) | 342
  Physical - Change at Cycle 7 | -4.62 (16.23)
  Physical - Change at Cycle 9: number analyzed (Participants) | 275
  Physical - Change at Cycle 9 | -4.36 (15.79)
  Physical - Change at Cycle 11: number analyzed (Participants) | 235
  Physical - Change at Cycle 11 | -6.99 (17.89)
  Physical - Change at Cycle 13: number analyzed (Participants) | 154
  Physical - Change at Cycle 13 | -4.99 (16.17)
  Physical - Change at Cycle 15: number analyzed (Participants) | 122
  Physical - Change at Cycle 15 | -3.54 (15.99)
  Physical - Change at Cycle 17: number analyzed (Participants) | 87
  Physical - Change at Cycle 17 | -5.10 (16.20)
  Physical - Change at Cycle 19: number analyzed (Participants) | 61
  Physical - Change at Cycle 19 | -5.68 (16.23)
  Physical - Change at Cycle 21: number analyzed (Participants) | 46
  Physical - Change at Cycle 21 | -5.70 (13.01)
  Physical - Change at Cycle 23: number analyzed (Participants) | 36
  Physical - Change at Cycle 23 | -7.87 (14.38)
  Physical - Change at Cycle 25: number analyzed (Participants) | 29
  Physical - Change at Cycle 25 | -5.75 (12.18)
  Physical - Change at Cycle 27: number analyzed (Participants) | 23
  Physical - Change at Cycle 27 | -6.59 (11.64)
  Physical - Change at Cycle 29: number analyzed (Participants) | 20
  Physical - Change at Cycle 29 | -7.67 (11.09)
  Physical - Change at Cycle 31: number analyzed (Participants) | 15
  Physical - Change at Cycle 31 | -9.33 (14.65)
  Physical - Change at Cycle 33: number analyzed (Participants) | 11
  Physical - Change at Cycle 33 | -5.45 (9.81)
  Physical - Change at Cycle 35: number analyzed (Participants) | 10
  Physical - Change at Cycle 35 | -10.00 (13.05)
  Physical - Change at EOT: number analyzed (Participants) | 341
  Physical - Change at EOT | -11.16 (21.65)
  Role - Baseline: number analyzed (Participants) | 633
  Role - Baseline | 79.91 (26.25)
  Role - Change at Cycle 3: number analyzed (Participants) | 551
  Role - Change at Cycle 3 | -6.26 (25.22)
  Role - Change at Cycle 5: number analyzed (Participants) | 442
  Role - Change at Cycle 5 | -5.66 (23.26)
  Role - Change at Cycle 7: number analyzed (Participants) | 342
  Role - Change at Cycle 7 | -6.68 (24.29)
  Role - Change at Cycle 9: number analyzed (Participants) | 275
  Role - Change at Cycle 9 | -6.55 (23.95)
  Role - Change at Cycle 11: number analyzed (Participants) | 234
  Role - Change at Cycle 11 | -8.76 (26.35)
  Role - Change at Cycle 13: number analyzed (Participants) | 154
  Role - Change at Cycle 13 | -7.36 (23.41)
  Role - Change at Cycle 15: number analyzed (Participants) | 123
  Role - Change at Cycle 15 | -7.18 (21.98)
  Role - Change at Cycle 17: number analyzed (Participants) | 87
  Role - Change at Cycle 17 | -9.58 (22.54)
  Role - Change at Cycle 19: number analyzed (Participants) | 61
  Role - Change at Cycle 19 | -9.84 (22.44)
  Role - Change at Cycle 21: number analyzed (Participants) | 46
  Role - Change at Cycle 21 | -9.78 (18.11)
  Role - Change at Cycle 23: number analyzed (Participants) | 36
  Role - Change at Cycle 23 | -10.65 (18.32)
  Role - Change at Cycle 25: number analyzed (Participants) | 29
  Role - Change at Cycle 25 | -10.92 (17.97)
  Role - Change at Cycle 27: number analyzed (Participants) | 23
  Role - Change at Cycle 27 | -10.14 (17.22)
  Role - Change at Cycle 29: number analyzed (Participants) | 20
  Role - Change at Cycle 29 | -10.83 (17.33)
  Role - Change at Cycle 31: number analyzed (Participants) | 15
  Role - Change at Cycle 31 | -14.44 (18.76)
  Role - Change at Cycle 33: number analyzed (Participants) | 11
  Role - Change at Cycle 33 | -15.15 (15.73)
  Role - Change at Cycle 35: number analyzed (Participants) | 10
  Role - Change at Cycle 35 | -15.00 (16.57)
  Role - Change at EOT: number analyzed (Participants) | 340
  Role - Change at EOT | -12.11 (28.22)
  Emotional - Baseline: number analyzed (Participants) | 634
  Emotional - Baseline | 78.96 (20.60)
  Emotional - Change at Cycle 3: number analyzed (Participants) | 553
  Emotional - Change at Cycle 3 | 1.14 (19.95)
  Emotional - Change at Cycle 5: number analyzed (Participants) | 436
  Emotional - Change at Cycle 5 | 0.74 (19.32)
  Emotional - Change at Cycle 7: number analyzed (Participants) | 344
  Emotional - Change at Cycle 7 | 1.58 (20.91)
  Emotional - Change at Cycle 9: number analyzed (Participants) | 275
  Emotional - Change at Cycle 9 | 1.69 (21.38)
  Emotional - Change at Cycle 11: number analyzed (Participants) | 235
  Emotional - Change at Cycle 11 | 0.08 (20.40)
  Emotional - Change at Cycle 13: number analyzed (Participants) | 152
  Emotional - Change at Cycle 13 | 0.93 (20.08)
  Emotional - Change at Cycle 15: number analyzed (Participants) | 124
  Emotional - Change at Cycle 15 | 2.51 (20.23)
  Emotional - Change at Cycle 17: number analyzed (Participants) | 87
  Emotional - Change at Cycle 17 | 2.91 (18.23)
  Emotional - Change at Cycle 19: number analyzed (Participants) | 60
  Emotional - Change at Cycle 19 | 1.39 (17.60)
  Emotional - Change at Cycle 21: number analyzed (Participants) | 44
  Emotional - Change at Cycle 21 | 0.06 (17.86)
  Emotional - Change at Cycle 23: number analyzed (Participants) | 35
  Emotional - Change at Cycle 23 | 1.75 (19.29)
  Emotional - Change at Cycle 25: number analyzed (Participants) | 29
  Emotional - Change at Cycle 25 | 4.98 (15.86)
  Emotional - Change at Cycle 27: number analyzed (Participants) | 23
  Emotional - Change at Cycle 27 | 1.57 (17.64)
  Emotional - Change at Cycle 29: number analyzed (Participants) | 20
  Emotional - Change at Cycle 29 | 2.64 (17.88)
  Emotional - Change at Cycle 31: number analyzed (Participants) | 15
  Emotional - Change at Cycle 31 | 1.30 (17.78)
  Emotional - Change at Cycle 33: number analyzed (Participants) | 11
  Emotional - Change at Cycle 33 | 0.25 (3.82)
  Emotional - Change at Cycle 35: number analyzed (Participants) | 10
  Emotional - Change at Cycle 35 | -0.00 (5.56)
  Emotional - Change at EOT: number analyzed (Participants) | 345
  Emotional - Change at EOT | -2.87 (22.52)
  Cognitive - Baseline: number analyzed (Participants) | 635
  Cognitive - Baseline | 86.90 (19.26)
  Cognitive - Change at Cycle 3: number analyzed (Participants) | 555
  Cognitive - Change at Cycle 3 | -1.77 (16.92)
  Cognitive - Change at Cycle 5: number analyzed (Participants) | 437
  Cognitive - Change at Cycle 5 | -1.87 (16.58)
  Cognitive - Change at Cycle 7: number analyzed (Participants) | 343
  Cognitive - Change at Cycle 7 | -1.99 (19.71)
  Cognitive - Change at Cycle 9: number analyzed (Participants) | 275
  Cognitive - Change at Cycle 9 | -2.18 (20.17)
  Cognitive - Change at Cycle 11: number analyzed (Participants) | 234
  Cognitive - Change at Cycle 11 | -4.27 (20.29)
  Cognitive - Change at Cycle 13: number analyzed (Participants) | 153
  Cognitive - Change at Cycle 13 | -2.83 (17.40)
  Cognitive - Change at Cycle 15: number analyzed (Participants) | 124
  Cognitive - Change at Cycle 15 | -2.28 (19.40)
  Cognitive - Change at Cycle 17: number analyzed (Participants) | 87
  Cognitive - Change at Cycle 17 | -3.45 (19.38)
  Cognitive - Change at Cycle 19: number analyzed (Participants) | 60
  Cognitive - Change at Cycle 19 | -5.00 (22.19)
  Cognitive - Change at Cycle 21: number analyzed (Participants) | 45
  Cognitive - Change at Cycle 21 | -5.56 (16.28)
  Cognitive - Change at Cycle 23: number analyzed (Participants) | 35
  Cognitive - Change at Cycle 23 | -5.71 (14.54)
  Cognitive - Change at Cycle 25: number analyzed (Participants) | 29
  Cognitive - Change at Cycle 25 | -6.90 (21.14)
  Cognitive - Change at Cycle 27: number analyzed (Participants) | 23
  Cognitive - Change at Cycle 27 | -5.80 (16.37)
  Cognitive - Change at Cycle 29: number analyzed (Participants) | 20
  Cognitive - Change at Cycle 29 | -6.67 (18.26)
  Cognitive - Change at Cycle 31: number analyzed (Participants) | 15
  Cognitive - Change at Cycle 31 | -5.56 (15.00)
  Cognitive - Change at Cycle 33: number analyzed (Participants) | 11
  Cognitive - Change at Cycle 33 | -10.61 (17.12)
  Cognitive - Change at Cycle 35: number analyzed (Participants) | 10
  Cognitive - Change at Cycle 35 | -11.67 (13.72)
  Cognitive- Change at EOT: number analyzed (Participants) | 345
  Cognitive- Change at EOT | -4.98 (22.67)
  Social - Baseline: number analyzed (Participants) | 634
  Social - Baseline | 80.57 (24.68)
  Social - Change at Cycle 3: number analyzed (Participants) | 554
  Social - Change at Cycle 3 | -2.05 (22.83)
  Social - Change at Cycle 5: number analyzed (Participants) | 437
  Social - Change at Cycle 5 | -2.86 (21.60)
  Social - Change at Cycle 7: number analyzed (Participants) | 345
  Social - Change at Cycle 7 | -4.78 (23.65)
  Social - Change at Cycle 9: number analyzed (Participants) | 274
  Social - Change at Cycle 9 | -4.56 (23.84)
  Social - Change at Cycle 11: number analyzed (Participants) | 235
  Social - Change at Cycle 11 | -7.09 (24.83)
  Social - Change at Cycle 13: number analyzed (Participants) | 153
  Social - Change at Cycle 13 | -5.56 (24.03)
  Social - Change at Cycle 15: number analyzed (Participants) | 124
  Social - Change at Cycle 15 | -6.18 (23.23)
  Social - Change at Cycle 17: number analyzed (Participants) | 87
  Social - Change at Cycle 17 | -5.56 (22.69)
  Social - Change at Cycle 19: number analyzed (Participants) | 60
  Social - Change at Cycle 19 | -5.28 (22.02)
  Social - Change at Cycle 21: number analyzed (Participants) | 45
  Social - Change at Cycle 21 | -5.56 (21.61)
  Social - Change at Cycle 23: number analyzed (Participants) | 35
  Social - Change at Cycle 23 | -7.62 (17.78)
  Social - Change at Cycle 25: number analyzed (Participants) | 29
  Social - Change at Cycle 25 | -4.60 (18.31)
  Social - Change at Cycle 27: number analyzed (Participants) | 23
  Social - Change at Cycle 27 | -2.17 (17.63)
  Social - Change at Cycle 29: number analyzed (Participants) | 20
  Social - Change at Cycle 29 | -5.00 (18.81)
  Social - Change at Cycle 31: number analyzed (Participants) | 15
  Social - Change at Cycle 31 | -7.78 (25.09)
  Social - Change at Cycle 33: number analyzed (Participants) | 11
  Social - Change at Cycle 33 | -1.52 (17.41)
  Social - Change at Cycle 35: number analyzed (Participants) | 10
  Social - Change at Cycle 35 | -1.67 (14.59)
  Social - Change at EOT: number analyzed (Participants) | 344
  Social - Change at EOT | -9.01 (26.23)

16. Secondary Outcome: Change From Baseline in HRQL EORTC QLQ-C30 Score: Symptom Scales
Description: EORTC-QLQ-C30 is a cancer-specific instrument with 30 questions for evaluation of new chemotherapy and provides an assessment of participant reported outcome dimensions. First 28 questions used 4-point scale (1=not at all,2=a little,3=quite a bit,4=very much) for evaluating 5 functional scales (physical,role,emotional,cognitive,social), 3 symptom scales (fatigue,nausea/vomiting,pain) & other single items. For each item,high score represented high level of symptomatology/problem. Last 2 questions represented participant's assessment of overall health & quality of life, coded on 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 observed values and change from baseline for global health status (scoring of questions 29 & 30) and 5 functional scales, 3 symptom scales and other single items (scoring of questions 1 to 28). Answers were converted into grading scale, with values between 0 and 100. A high score represented a favorable outcome with a best quality of life for participant.
Time Frame: as for outcome 15
Population: EORTC QLQ-C30 analysis population. Here, "Number Analyzed = participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 636
units on a scale
  Fatigue - Baseline: number analyzed (Participants) | 633
  Fatigue - Baseline | 29.16 (23.48)
  Fatigue - Change at Cycle 3: number analyzed (Participants) | 551
  Fatigue - Change at Cycle 3 | 7.35 (21.62)
  Fatigue - Change at Cycle 5: number analyzed (Participants) | 443
  Fatigue - Change at Cycle 5 | 8.40 (21.88)
  Fatigue - Change at Cycle 7: number analyzed (Participants) | 344
  Fatigue - Change at Cycle 7 | 9.54 (22.60)
  Fatigue - Change at Cycle 9: number analyzed (Participants) | 276
  Fatigue - Change at Cycle 9 | 7.89 (21.80)
  Fatigue - Change at Cycle 11: number analyzed (Participants) | 235
  Fatigue - Change at Cycle 11 | 11.30 (23.73)
  Fatigue - Change at Cycle 13: number analyzed (Participants) | 154
  Fatigue - Change at Cycle 13 | 8.33 (21.72)
  Fatigue - Change at Cycle 15: number analyzed (Participants) | 123
  Fatigue - Change at Cycle 15 | 7.41 (22.38)
  Fatigue - Change at Cycle 17: number analyzed (Participants) | 87
  Fatigue - Change at Cycle 17 | 6.70 (21.25)
  Fatigue - Change at Cycle 19: number analyzed (Participants) | 61
  Fatigue - Change at Cycle 19 | 8.93 (19.83)
  Fatigue - Change at Cycle 21: number analyzed (Participants) | 46
  Fatigue - Change at Cycle 21 | 10.39 (17.90)
  Fatigue - Change at Cycle 23: number analyzed (Participants) | 36
  Fatigue - Change at Cycle 23 | 10.80 (18.49)
  Fatigue - Change at Cycle 25: number analyzed (Participants) | 29
  Fatigue - Change at Cycle 25 | 7.66 (19.94)
  Fatigue - Change at Cycle 27: number analyzed (Participants) | 23
  Fatigue - Change at Cycle 27 | 9.66 (18.74)
  Fatigue - Change at Cycle 29: number analyzed (Participants) | 20
  Fatigue - Change at Cycle 29 | 11.67 (18.55)
  Fatigue - Change at Cycle 31: number analyzed (Participants) | 15
  Fatigue - Change at Cycle 31 | 14.07 (21.61)
  Fatigue - Change at Cycle 33: number analyzed (Participants) | 11
  Fatigue - Change at Cycle 33 | 15.15 (21.81)
  Fatigue - Change at Cycle 35: number analyzed (Participants) | 10
  Fatigue - Change at Cycle 35 | 14.44 (18.92)
  Fatigue - Change at EOT: number analyzed (Participants) | 343
  Fatigue - Change at EOT | 12.31 (25.56)
  Nausea and Vomiting - Baseline: number analyzed (Participants) | 635
  Nausea and Vomiting - Baseline | 5.88 (13.99)
  Nausea and Vomiting - Change at Cycle 3: number analyzed (Participants) | 554
  Nausea and Vomiting - Change at Cycle 3 | 6.68 (19.81)
  Nausea and Vomiting - Change at Cycle 5: number analyzed (Participants) | 442
  Nausea and Vomiting - Change at Cycle 5 | 6.98 (19.79)
  Nausea and Vomiting - Change at Cycle 7: number analyzed (Participants) | 343
  Nausea and Vomiting - Change at Cycle 7 | 6.61 (18.07)
  Nausea and Vomiting - Change at Cycle 9: number analyzed (Participants) | 277
  Nausea and Vomiting - Change at Cycle 9 | 6.20 (19.68)
  Nausea and Vomiting - Change at Cycle 11: number analyzed (Participants) | 236
  Nausea and Vomiting - Change at Cycle 11 | 8.97 (19.83)
  Nausea and Vomiting - Change at Cycle 13: number analyzed (Participants) | 154
  Nausea and Vomiting - Change at Cycle 13 | 6.82 (14.71)
  Nausea and Vomiting - Change at Cycle 15: number analyzed (Participants) | 124
  Nausea and Vomiting - Change at Cycle 15 | 6.85 (16.33)
  Nausea and Vomiting - Change at Cycle 17: number analyzed (Participants) | 87
  Nausea and Vomiting - Change at Cycle 17 | 3.45 (15.49)
  Nausea and Vomiting - Change at Cycle 19: number analyzed (Participants) | 61
  Nausea and Vomiting - Change at Cycle 19 | 6.56 (14.04)
  Nausea and Vomiting - Change at Cycle 21: number analyzed (Participants) | 46
  Nausea and Vomiting - Change at Cycle 21 | 3.99 (14.14)
  Nausea and Vomiting - Change at Cycle 23: number analyzed (Participants) | 36
  Nausea and Vomiting - Change at Cycle 23 | 7.87 (10.90)
  Nausea and Vomiting - Change at Cycle 25: number analyzed (Participants) | 29
  Nausea and Vomiting - Change at Cycle 25 | 4.02 (8.52)
  Nausea and Vomiting - Change at Cycle 27: number analyzed (Participants) | 23
  Nausea and Vomiting - Change at Cycle 27 | 7.25 (11.04)
  Nausea and Vomiting - Change at Cycle 29: number analyzed (Participants) | 20
  Nausea and Vomiting - Change at Cycle 29 | 1.67 (5.13)
  Nausea and Vomiting - Change at Cycle 31: number analyzed (Participants) | 15
  Nausea and Vomiting - Change at Cycle 31 | 13.33 (28.31)
  Nausea and Vomiting - Change at Cycle 33: number analyzed (Participants) | 11
  Nausea and Vomiting - Change at Cycle 33 | 3.03 (6.74)
  Nausea and Vomiting - Change at Cycle 35: number analyzed (Participants) | 10
  Nausea and Vomiting - Change at Cycle 35 | 3.33 (7.03)
  Nausea and Vomiting - Change at EOT: number analyzed (Participants) | 344
  Nausea and Vomiting - Change at EOT | 6.64 (21.11)
  Pain - Baseline | 20.47 (25.08)
  Pain - Change at Cycle 3: number analyzed (Participants) | 554
  Pain - Change at Cycle 3 | 2.68 (25.02)
  Pain - Change at Cycle 5: number analyzed (Participants) | 444
  Pain - Change at Cycle 5 | 2.52 (23.48)
  Pain - Change at Cycle 7: number analyzed (Participants) | 345
  Pain - Change at Cycle 7 | 3.00 (24.98)
  Pain - Change at Cycle 9: number analyzed (Participants) | 276
  Pain - Change at Cycle 9 | 2.72 (24.45)
  Pain - Change at Cycle 11: number analyzed (Participants) | 236
  Pain - Change at Cycle 11 | 6.64 (23.68)
  Pain - Change at Cycle 13: number analyzed (Participants) | 155
  Pain - Change at Cycle 13 | 5.16 (19.79)
  Pain - Change at Cycle 15: number analyzed (Participants) | 124
  Pain - Change at Cycle 15 | 7.26 (21.91)
  Pain - Change at Cycle 17: number analyzed (Participants) | 87
  Pain - Change at Cycle 17 | 9.39 (22.97)
  Pain - Change at Cycle 19: number analyzed (Participants) | 61
  Pain - Change at Cycle 19 | 8.74 (22.28)
  Pain - Change at Cycle 21: number analyzed (Participants) | 46
  Pain - Change at Cycle 21 | 7.25 (18.14)
  Pain - Change at Cycle 23: number analyzed (Participants) | 36
  Pain - Change at Cycle 23 | 8.33 (19.31)
  Pain - Change at Cycle 25: number analyzed (Participants) | 29
  Pain - Change at Cycle 25 | 5.75 (21.02)
  Pain - Change at Cycle 27: number analyzed (Participants) | 23
  Pain - Change at Cycle 27 | 5.07 (17.72)
  Pain - Change at Cycle 29: number analyzed (Participants) | 20
  Pain - Change at Cycle 29 | 4.17 (16.11)
  Pain - Change at Cycle 31: number analyzed (Participants) | 15
  Pain - Change at Cycle 31 | 10.00 (23.40)
  Pain - Change at Cycle 33: number analyzed (Participants) | 11
  Pain - Change at Cycle 33 | 7.58 (22.81)
  Pain - Change at Cycle 35: number analyzed (Participants) | 10
  Pain - Change at Cycle 35 | 6.67 (21.08)
  Pain - Change at EOT: number analyzed (Participants) | 347
  Pain - Change at EOT | 10.85 (28.99)
  Dyspnoea - Baseline: number analyzed (Participants) | 627
  Dyspnoea - Baseline | 13.45 (22.01)
  Dyspnoea - Change at Cycle 3: number analyzed (Participants) | 542
  Dyspnoea - Change at Cycle 3 | 3.63 (22.96)
  Dyspnoea - Change at Cycle 5: number analyzed (Participants) | 435
  Dyspnoea - Change at Cycle 5 | 5.75 (24.06)
  Dyspnoea - Change at Cycle 7: number analyzed (Participants) | 339
  Dyspnoea - Change at Cycle 7 | 6.98 (24.47)
  Dyspnoea - Change at Cycle 9: number analyzed (Participants) | 271
  Dyspnoea - Change at Cycle 9 | 6.89 (24.38)
  Dyspnoea - Change at Cycle 11: number analyzed (Participants) | 232
  Dyspnoea - Change at Cycle 11 | 8.19 (26.59)
  Dyspnoea - Change at Cycle 13: number analyzed (Participants) | 152
  Dyspnoea - Change at Cycle 13 | 6.36 (25.37)
  Dyspnoea - Change at Cycle 15: number analyzed (Participants) | 121
  Dyspnoea - Change at Cycle 15 | 3.58 (24.65)
  Dyspnoea - Change at Cycle 17: number analyzed (Participants) | 84
  Dyspnoea - Change at Cycle 17 | 5.16 (24.54)
  Dyspnoea - Change at Cycle 19: number analyzed (Participants) | 59
  Dyspnoea - Change at Cycle 19 | 6.78 (26.82)
  Dyspnoea - Change at Cycle 21: number analyzed (Participants) | 44
  Dyspnoea - Change at Cycle 21 | 3.79 (22.98)
  Dyspnoea - Change at Cycle 23: number analyzed (Participants) | 33
  Dyspnoea - Change at Cycle 23 | 4.04 (20.00)
  Dyspnoea - Change at Cycle 25: number analyzed (Participants) | 27
  Dyspnoea - Change at Cycle 25 | 1.23 (21.64)
  Dyspnoea - Change at Cycle 27: number analyzed (Participants) | 22
  Dyspnoea - Change at Cycle 27 | 3.03 (22.79)
  Dyspnoea - Change at Cycle 29: number analyzed (Participants) | 19
  Dyspnoea - Change at Cycle 29 | -1.75 (23.50)
  Dyspnoea - Change at Cycle 31: number analyzed (Participants) | 14
  Dyspnoea - Change at Cycle 31 | 16.67 (28.50)
  Dyspnoea - Change at Cycle 33: number analyzed (Participants) | 10
  Dyspnoea - Change at Cycle 33 | 16.67 (17.57)
  Dyspnoea - Change at Cycle 35: number analyzed (Participants) | 10
  Dyspnoea - Change at Cycle 35 | 16.67 (23.57)
  Dyspnoea - Change at EOT: number analyzed (Participants) | 337
  Dyspnoea - Change at EOT | 6.53 (25.79)
  Insomnia - Baseline: number analyzed (Participants) | 628
  Insomnia - Baseline | 24.15 (28.09)
  Insomnia - Change at Cycle 3: number analyzed (Participants) | 544
  Insomnia - Change at Cycle 3 | 0.37 (27.36)
  Insomnia - Change at Cycle 5: number analyzed (Participants) | 438
  Insomnia - Change at Cycle 5 | -0.08 (28.48)
  Insomnia - Change at Cycle 7: number analyzed (Participants) | 338
  Insomnia - Change at Cycle 7 | -2.37 (29.63)
  Insomnia - Change at Cycle 9: number analyzed (Participants) | 274
  Insomnia - Change at Cycle 9 | -0.24 (29.37)
  Insomnia - Change at Cycle 11: number analyzed (Participants) | 234
  Insomnia - Change at Cycle 11 | 2.56 (28.86)
  Insomnia - Change at Cycle 13: number analyzed (Participants) | 153
  Insomnia - Change at Cycle 13 | 0.65 (26.89)
  Insomnia - Change at Cycle 15: number analyzed (Participants) | 122
  Insomnia - Change at Cycle 15 | -2.19 (27.01)
  Insomnia - Change at Cycle 17: number analyzed (Participants) | 87
  Insomnia - Change at Cycle 17 | -1.92 (25.60)
  Insomnia - Change at Cycle 19: number analyzed (Participants) | 61
  Insomnia - Change at Cycle 19 | 1.64 (23.12)
  Insomnia - Change at Cycle 21: number analyzed (Participants) | 45
  Insomnia - Change at Cycle 21 | 0.74 (25.11)
  Insomnia - Change at Cycle 23: number analyzed (Participants) | 36
  Insomnia - Change at Cycle 23 | -0.93 (33.32)
  Insomnia - Change at Cycle 25: number analyzed (Participants) | 29
  Insomnia - Change at Cycle 25 | -0.00 (28.17)
  Insomnia - Change at Cycle 27: number analyzed (Participants) | 22
  Insomnia - Change at Cycle 27 | -1.52 (24.07)
  Insomnia - Change at Cycle 29: number analyzed (Participants) | 20
  Insomnia - Change at Cycle 29 | -3.33 (30.40)
  Insomnia - Change at Cycle 31: number analyzed (Participants) | 15
  Insomnia - Change at Cycle 31 | -4.44 (41.53)
  Insomnia - Change at Cycle 33: number analyzed (Participants) | 11
  Insomnia - Change at Cycle 33 | -6.06 (32.72)
  Insomnia - Change at Cycle 35: number analyzed (Participants) | 10
  Insomnia - Change at Cycle 35 | -3.33 (33.15)
  Insomnia - Change at EOT: number analyzed (Participants) | 339
  Insomnia - Change at EOT | 5.31 (32.50)
  Appetite loss - Baseline: number analyzed (Participants) | 631
  Appetite loss - Baseline | 17.38 (26.01)
  Appetite loss - Change at Cycle 3: number analyzed (Participants) | 546
  Appetite loss - Change at Cycle 3 | 9.10 (28.64)
  Appetite loss - Change at Cycle 5: number analyzed (Participants) | 436
  Appetite loss - Change at Cycle 5 | 9.02 (28.14)
  Appetite loss - Change at Cycle 7: number analyzed (Participants) | 342
  Appetite loss - Change at Cycle 7 | 9.84 (27.80)
  Appetite loss - Change at Cycle 9: number analyzed (Participants) | 274
  Appetite loss - Change at Cycle 9 | 9.98 (27.18)
  Appetite loss - Change at Cycle 11: number analyzed (Participants) | 234
  Appetite loss - Change at Cycle 11 | 14.53 (28.27)
  Appetite loss - Change at Cycle 13: number analyzed (Participants) | 150
  Appetite loss - Change at Cycle 13 | 10.67 (27.12)
  Appetite loss - Change at Cycle 15: number analyzed (Participants) | 121
  Appetite loss - Change at Cycle 15 | 10.74 (25.90)
  Appetite loss - Change at Cycle 17: number analyzed (Participants) | 86
  Appetite loss - Change at Cycle 17 | 8.91 (24.75)
  Appetite loss - Change at Cycle 19: number analyzed (Participants) | 61
  Appetite loss - Change at Cycle 19 | 9.84 (24.60)
  Appetite loss - Change at Cycle 21: number analyzed (Participants) | 46
  Appetite loss - Change at Cycle 21 | 13.04 (25.80)
  Appetite loss - Change at Cycle 23: number analyzed (Participants) | 35
  Appetite loss - Change at Cycle 23 | 12.38 (25.67)
  Appetite loss - Change at Cycle 25: number analyzed (Participants) | 29
  Appetite loss - Change at Cycle 25 | 11.49 (20.46)
  Appetite loss - Change at Cycle 27: number analyzed (Participants) | 23
  Appetite loss - Change at Cycle 27 | 15.94 (22.18)
  Appetite loss - Change at Cycle 29: number analyzed (Participants) | 20
  Appetite loss - Change at Cycle 29 | 15.00 (20.16)
  Appetite loss - Change at Cycle 31: number analyzed (Participants) | 15
  Appetite loss - Change at Cycle 31 | 15.56 (24.77)
  Appetite loss - Change at Cycle 33: number analyzed (Participants) | 11
  Appetite loss - Change at Cycle 33 | 15.15 (22.92)
  Appetite loss - Change at Cycle 35: number analyzed (Participants) | 10
  Appetite loss - Change at Cycle 35 | 16.67 (17.57)
  Appetite loss - Change at EOT: number analyzed (Participants) | 338
  Appetite loss - Change at EOT | 12.03 (33.48)
  Constipation - Baseline: number analyzed (Participants) | 632
  Constipation - Baseline | 12.71 (21.61)
  Constipation - Change at Cycle 3: number analyzed (Participants) | 550
  Constipation - Change at Cycle 3 | 2.42 (25.25)
  Constipation - Change at Cycle 5: number analyzed (Participants) | 433
  Constipation - Change at Cycle 5 | 3.77 (26.52)
  Constipation - Change at Cycle 7: number analyzed (Participants) | 342
  Constipation - Change at Cycle 7 | 2.63 (26.09)
  Constipation - Change at Cycle 9: number analyzed (Participants) | 274
  Constipation - Change at Cycle 9 | 5.35 (26.68)
  Constipation - Change at Cycle 11: number analyzed (Participants) | 234
  Constipation - Change at Cycle 11 | 4.42 (26.47)
  Constipation - Change at Cycle 13: number analyzed (Participants) | 153
  Constipation - Change at Cycle 13 | 4.58 (25.95)
  Constipation - Change at Cycle 15: number analyzed (Participants) | 122
  Constipation - Change at Cycle 15 | 4.92 (26.30)
  Constipation - Change at Cycle 17: number analyzed (Participants) | 86
  Constipation - Change at Cycle 17 | 5.43 (23.35)
  Constipation - Change at Cycle 19: number analyzed (Participants) | 60
  Constipation - Change at Cycle 19 | 8.33 (21.81)
  Constipation - Change at Cycle 21: number analyzed (Participants) | 44
  Constipation - Change at Cycle 21 | 6.06 (18.00)
  Constipation - Change at Cycle 23: number analyzed (Participants) | 36
  Constipation - Change at Cycle 23 | 9.26 (21.98)
  Constipation - Change at Cycle 25: number analyzed (Participants) | 29
  Constipation - Change at Cycle 25 | 5.75 (17.97)
  Constipation - Change at Cycle 27: number analyzed (Participants) | 23
  Constipation - Change at Cycle 27 | 1.45 (12.22)
  Constipation - Change at Cycle 29: number analyzed (Participants) | 20
  Constipation - Change at Cycle 29 | 6.67 (20.52)
  Constipation - Change at Cycle 31: number analyzed (Participants) | 15
  Constipation - Change at Cycle 31 | 22.22 (32.53)
  Constipation - Change at Cycle 33: number analyzed (Participants) | 11
  Constipation - Change at Cycle 33 | 12.12 (16.82)
  Constipation - Change at Cycle 35: number analyzed (Participants) | 10
  Constipation - Change at Cycle 35 | 10.00 (16.10)
  Constipation - Change at EOT: number analyzed (Participants) | 344
  Constipation - Change at EOT | 3.78 (27.33)
  Diarrhoea - Baseline: number analyzed (Participants) | 633
  Diarrhoea - Baseline | 10.37 (19.47)
  Diarrhoea - Change at Cycle 3: number analyzed (Participants) | 549
  Diarrhoea - Change at Cycle 3 | 11.72 (28.16)
  Diarrhoea - Change at Cycle 5: number analyzed (Participants) | 433
  Diarrhoea - Change at Cycle 5 | 10.85 (28.29)
  Diarrhoea - Change at Cycle 7: number analyzed (Participants) | 344
  Diarrhoea - Change at Cycle 7 | 14.63 (29.94)
  Diarrhoea - Change at Cycle 9: number analyzed (Participants) | 274
  Diarrhoea - Change at Cycle 9 | 11.44 (26.44)
  Diarrhoea - Change at Cycle 11: number analyzed (Participants) | 235
  Diarrhoea - Change at Cycle 11 | 15.46 (27.26)
  Diarrhoea - Change at Cycle 13: number analyzed (Participants) | 151
  Diarrhoea - Change at Cycle 13 | 11.26 (24.00)
  Diarrhoea - Change at Cycle 15: number analyzed (Participants) | 121
  Diarrhoea - Change at Cycle 15 | 11.02 (28.02)
  Diarrhoea - Change at Cycle 17: number analyzed (Participants) | 87
  Diarrhoea - Change at Cycle 17 | 10.34 (21.75)
  Diarrhoea - Change at Cycle 19: number analyzed (Participants) | 59
  Diarrhoea - Change at Cycle 19 | 15.25 (25.76)
  Diarrhoea - Change at Cycle 21: number analyzed (Participants) | 45
  Diarrhoea - Change at Cycle 21 | 14.07 (24.09)
  Diarrhoea - Change at Cycle 23: number analyzed (Participants) | 36
  Diarrhoea - Change at Cycle 23 | 18.52 (21.74)
  Diarrhoea - Change at Cycle 25: number analyzed (Participants) | 29
  Diarrhoea - Change at Cycle 25 | 10.34 (22.01)
  Diarrhoea - Change at Cycle 27: number analyzed (Participants) | 22
  Diarrhoea - Change at Cycle 27 | 13.64 (19.68)
  Diarrhoea - Change at Cycle 29: number analyzed (Participants) | 20
  Diarrhoea - Change at Cycle 29 | 16.67 (25.36)
  Diarrhoea - Change at Cycle 31: number analyzed (Participants) | 15
  Diarrhoea - Change at Cycle 31 | 20.00 (24.56)
  Diarrhoea - Change at Cycle 33: number analyzed (Participants) | 11
  Diarrhoea - Change at Cycle 33 | 18.18 (22.92)
  Diarrhoea - Change at Cycle 35: number analyzed (Participants) | 10
  Diarrhoea - Change at Cycle 35 | 30.00 (18.92)
  Diarrhoea - Change at EOT: number analyzed (Participants) | 342
  Diarrhoea - Change at EOT | 7.31 (24.26)
  Financial difficulties - Baseline: number analyzed (Participants) | 628
  Financial difficulties - Baseline | 20.12 (30.25)
  Financial difficulties - Change at Cycle 3: number analyzed (Participants) | 547
  Financial difficulties - Change at Cycle 3 | -1.83 (23.80)
  Financial difficulties - Change at Cycle 5: number analyzed (Participants) | 430
  Financial difficulties - Change at Cycle 5 | -1.32 (24.00)
  Financial difficulties - Change at Cycle 7: number analyzed (Participants) | 337
  Financial difficulties - Change at Cycle 7 | -0.99 (27.68)
  Financial difficulties - Change at Cycle 9: number analyzed (Participants) | 270
  Financial difficulties - Change at Cycle 9 | -0.49 (26.80)
  Financial difficulties - Change at Cycle 11: number analyzed (Participants) | 232
  Financial difficulties - Change at Cycle 11 | 3.30 (25.64)
  Financial difficulties - Change at Cycle 13: number analyzed (Participants) | 150
  Financial difficulties - Change at Cycle 13 | 1.11 (27.96)
  Financial difficulties - Change at Cycle 15: number analyzed (Participants) | 122
  Financial difficulties - Change at Cycle 15 | -0.27 (27.94)
  Financial difficulties - Change at Cycle 17: number analyzed (Participants) | 87
  Financial difficulties - Change at Cycle 17 | 0.77 (27.36)
  Financial difficulties - Change at Cycle 19: number analyzed (Participants) | 60
  Financial difficulties - Change at Cycle 19 | 1.67 (29.70)
  Financial difficulties - Change at Cycle 21: number analyzed (Participants) | 45
  Financial difficulties - Change at Cycle 21 | 4.44 (25.23)
  Financial difficulties - Change at Cycle 23: number analyzed (Participants) | 34
  Financial difficulties - Change at Cycle 23 | 2.94 (23.74)
  Financial difficulties - Change at Cycle 25: number analyzed (Participants) | 29
  Financial difficulties - Change at Cycle 25 | -4.60 (19.36)
  Financial difficulties - Change at Cycle 27: number analyzed (Participants) | 23
  Financial difficulties - Change at Cycle 27 | -2.90 (24.44)
  Financial difficulties - Change at Cycle 29: number analyzed (Participants) | 20
  Financial difficulties - Change at Cycle 29 | 0.00 (21.63)
  Financial difficulties - Change at Cycle 31: number analyzed (Participants) | 15
  Financial difficulties - Change at Cycle 31 | -2.22 (19.79)
  Financial difficulties - Change at Cycle 33: number analyzed (Participants) | 11
  Financial difficulties - Change at Cycle 33 | -3.03 (17.98)
  Financial difficulties - Change at Cycle 35: number analyzed (Participants) | 10
  Financial difficulties - Change at Cycle 35 | 0.00 (15.71)
  Financial difficulties - Change at EOT: number analyzed (Participants) | 337
  Financial difficulties - Change at EOT | 2.97 (27.90)

17. Secondary Outcome: Change From Baseline in HRQL EQ-5D-3L Quality of Life: Single Index Utility Score
Description: EQ-5D was a standardized HRQL questionnaire consisting of EQ-5D descriptive system and Visual Analogue Scale (VAS). EQ-5D descriptive system comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression measured on 3 levels (no problem, some problems & severe problems) within a particular EQ-5D dimension. 5 dimensional 3-level system was converted into single index utility score. Possible values for single index utility score ranged from -0.594 (severe problems in all dimensions) to 1.0 (no problem in all dimensions) on scale where 1 represented best possible health state.
Time Frame: as for outcome 15
Population: EQ-5D analysis population: participants who signed informed consent form, had an evaluable EQ-5D questionnaire at baseline and at least one evaluable assessment post baseline and received at least part of one dose of study treatment (either Aflibercept or FOLFIRI). Here, 'Number Analyzed' = participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 623
units on a scale
  Baseline | 0.77 (0.24)
  Change at Cycle 3: number analyzed (Participants) | 536
  Change at Cycle 3 | -0.02 (0.23)
  Change at Cycle 5: number analyzed (Participants) | 428
  Change at Cycle 5 | -0.03 (0.22)
  Change at Cycle 7: number analyzed (Participants) | 335
  Change at Cycle 7 | -0.04 (0.23)
  Change at Cycle 9: number analyzed (Participants) | 269
  Change at Cycle 9 | -0.05 (0.24)
  Change at Cycle 11: number analyzed (Participants) | 226
  Change at Cycle 11 | -0.07 (0.25)
  Change at Cycle 13: number analyzed (Participants) | 149
  Change at Cycle 13 | -0.05 (0.20)
  Change at Cycle 15: number analyzed (Participants) | 119
  Change at Cycle 15 | -0.06 (0.23)
  Change at Cycle 17: number analyzed (Participants) | 81
  Change at Cycle 17 | -0.05 (0.24)
  Change at Cycle 19: number analyzed (Participants) | 58
  Change at Cycle 19 | -0.05 (0.18)
  Change at Cycle 21: number analyzed (Participants) | 44
  Change at Cycle 21 | -0.09 (0.20)
  Change at Cycle 23: number analyzed (Participants) | 34
  Change at Cycle 23 | -0.14 (0.26)
  Change at Cycle 25: number analyzed (Participants) | 28
  Change at Cycle 25 | -0.08 (0.21)
  Change at Cycle 27: number analyzed (Participants) | 23
  Change at Cycle 27 | -0.08 (0.21)
  Change at Cycle 29: number analyzed (Participants) | 20
  Change at Cycle 29 | -0.08 (0.20)
  Change at Cycle 31: number analyzed (Participants) | 15
  Change at Cycle 31 | -0.12 (0.30)
  Change at Cycle 33: number analyzed (Participants) | 11
  Change at Cycle 33 | 0.02 (0.14)
  Change at Cycle 35: number analyzed (Participants) | 10
  Change at Cycle 35 | -0.05 (0.14)
  Change at EOT: number analyzed (Participants) | 343
  Change at EOT | -0.11 (0.30)

18. Secondary Outcome: Change From Baseline in HRQL EQ-5D-3L VAS Score
Description: EQ-5D was a standardized HRQL questionnaire consisting of EQ-5D descriptive system and VAS. EQ-5D descriptive system comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression measured on 3 levels (no problem, some problems & severe problems) within a particular EQ-5D dimension. 5 dimensional 3-level system was converted into single index utility score. The VAS recorded the respondent's self-rated health on a vertical visual analogue scale. The VAS 'thermometer' has endpoints of 100 (Best imaginable health state) at the top and 0 (Worst imaginable health state) at the bottom. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
Time Frame: as for outcome 15
Population: EQ-5D analysis population. Here, 'Number Analyzed' = participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
Number analyzed (Participants) | 623
units on a scale
  Baseline: number analyzed (Participants) | 577
  Baseline | 72.81 (18.28)
  Change at Cycle 3: number analyzed (Participants) | 482
  Change at Cycle 3 | -1.85 (15.35)
  Change at Cycle 5: number analyzed (Participants) | 381
  Change at Cycle 5 | -2.15 (14.31)
  Change at Cycle 7: number analyzed (Participants) | 303
  Change at Cycle 7 | -2.20 (16.33)
  Change at Cycle 9: number analyzed (Participants) | 236
  Change at Cycle 9 | -2.74 (14.28)
  Change at Cycle 11: number analyzed (Participants) | 203
  Change at Cycle 11 | -3.10 (14.40)
  Change at Cycle 13: number analyzed (Participants) | 134
  Change at Cycle 13 | -2.36 (15.29)
  Change at Cycle 15: number analyzed (Participants) | 103
  Change at Cycle 15 | -1.05 (15.51)
  Change at Cycle 17: number analyzed (Participants) | 74
  Change at Cycle 17 | -1.91 (13.54)
  Change at Cycle 19: number analyzed (Participants) | 52
  Change at Cycle 19 | -3.06 (13.85)
  Change at Cycle 21: number analyzed (Participants) | 38
  Change at Cycle 21 | -2.13 (14.98)
  Change at Cycle 23: number analyzed (Participants) | 30
  Change at Cycle 23 | -5.77 (13.50)
  Change at Cycle 25: number analyzed (Participants) | 25
  Change at Cycle 25 | -7.28 (10.53)
  Change at Cycle 27: number analyzed (Participants) | 17
  Change at Cycle 27 | -4.94 (8.68)
  Change at Cycle 29: number analyzed (Participants) | 15
  Change at Cycle 29 | -8.80 (10.12)
  Change at Cycle 31: number analyzed (Participants) | 13
  Change at Cycle 31 | -6.69 (12.61)
  Change at Cycle 33: number analyzed (Participants) | 10
  Change at Cycle 33 | -7.90 (13.08)
  Change at Cycle 35: number analyzed (Participants) | 8
  Change at Cycle 35 | -8.88 (11.53)
  Change at EOT: number analyzed (Participants) | 310
  Change at EOT | -6.67 (17.38)

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to the final visit (214 weeks) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment-emergent that is AEs that developed/worsened and deaths that occurred during 'on-treatment period' (from the first dose of treatment to 30 days after the last dose of treatment [either aflibercept or FOLFIRI]). Analysis was performed on safety population.
Arm/Group | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin)
All-Cause Mortality (participants affected / at risk) | 48/779
Serious Adverse Events (participants affected / at risk) | 272/779
Other Adverse Events (participants affected / at risk) | 744/779
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin) (N=779)
Anaemia (Blood and lymphatic system disorders) | 7
Febrile Neutropenia (Blood and lymphatic system disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 2
Angina Pectoris (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Atrial Flutter (Cardiac disorders) | 2
Atrial Thrombosis (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 1
Coronary Artery Thrombosis (Cardiac disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 2
Ventricular Tachycardia (Cardiac disorders) | 1
Retinal Detachment (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 8
Abdominal Pain Upper (Gastrointestinal disorders) | 4
Anal Fissure (Gastrointestinal disorders) | 1
Anal Fistula (Gastrointestinal disorders) | 1
Anorectal Ulcer (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 39
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 2
Enterocutaneous Fistula (Gastrointestinal disorders) | 4
Enterovesical Fistula (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Fistula Of Small Intestine (Gastrointestinal disorders) | 1
Gastrointestinal Fistula (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Haemorrhoids Thrombosed (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Ileus Paralytic (Gastrointestinal disorders) | 1
Inguinal Hernia (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 12
Intestinal Perforation (Gastrointestinal disorders) | 4
Large Intestine Perforation (Gastrointestinal disorders) | 4
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 2
Rectal Perforation (Gastrointestinal disorders) | 1
Rectal Tenesmus (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 9
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 2
Chest Pain (General disorders) | 1
Disease Progression (General disorders) | 23
Fatigue (General disorders) | 4
General Physical Health Deterioration (General disorders) | 5
Malaise (General disorders) | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 12
Sudden Death (General disorders) | 2
Cholangitis (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis Acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 1
Portal Hypertension (Hepatobiliary disorders) | 1
Anaphylactic Shock (Immune system disorders) | 1
Abdominal Abscess (Infections and infestations) | 2
Abdominal Infection (Infections and infestations) | 1
Abdominal Wall Abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Catheter Site Abscess (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 7
Diabetic Foot Infection (Infections and infestations) | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1
Febrile Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis Escherichia Coli (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Herpes Zoster Meningoencephalitis (Infections and infestations) | 1
Infection (Infections and infestations) | 5
Infective Myositis (Infections and infestations) | 1
Klebsiella Infection (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 3
Lung Infection (Infections and infestations) | 3
Neutropenic Infection (Infections and infestations) | 1
Neutropenic Sepsis (Infections and infestations) | 3
Parainfluenzae Virus Infection (Infections and infestations) | 1
Pelvic Abscess (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Phlebitis Infective (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Pyelonephritis (Infections and infestations) | 1
Rectal Abscess (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 7
Septic Shock (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Streptococcal Bacteraemia (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 2
Tuberculosis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 5
Urosepsis (Infections and infestations) | 1
Accidental Exposure To Product (Injury, poisoning and procedural complications) | 2
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Anastomotic Leak (Injury, poisoning and procedural complications) | 1
Contrast Media Reaction (Injury, poisoning and procedural complications) | 1
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1
Meniscus Injury (Injury, poisoning and procedural complications) | 1
Stoma Site Haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 3
Subarachnoid Haemorrhage (Nervous system disorders) | 1
White Matter Lesion (Nervous system disorders) | 1
Thrombosis In Device (Product Issues) | 1
Confusional State (Psychiatric disorders) | 4
Acute Kidney Injury (Renal and urinary disorders) | 3
Hydronephrosis (Renal and urinary disorders) | 3
Nephrotic Syndrome (Renal and urinary disorders) | 5
Prerenal Failure (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Urinary Retention (Renal and urinary disorders) | 2
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Thoracic Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cancer Surgery (Surgical and medical procedures) | 2
Deep Vein Thrombosis (Vascular disorders) | 4
Hypertension (Vascular disorders) | 11
Hypotension (Vascular disorders) | 2
Orthostatic Hypotension (Vascular disorders) | 1
Peripheral Ischaemia (Vascular disorders) | 1
Vena Cava Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + FOLFIRI (Irinotecan, 5-FU & Leucovorin) (N=779)
Neutropenia (Blood and lymphatic system disorders) | 277
Abdominal Pain (Gastrointestinal disorders) | 150
Abdominal Pain Upper (Gastrointestinal disorders) | 67
Constipation (Gastrointestinal disorders) | 148
Diarrhoea (Gastrointestinal disorders) | 464
Nausea (Gastrointestinal disorders) | 337
Proctalgia (Gastrointestinal disorders) | 39
Stomatitis (Gastrointestinal disorders) | 329
Vomiting (Gastrointestinal disorders) | 190
Asthenia (General disorders) | 192
Fatigue (General disorders) | 283
Pyrexia (General disorders) | 87
Weight Decreased (Investigations) | 171
Decreased Appetite (Metabolism and nutrition disorders) | 206
Back Pain (Musculoskeletal and connective tissue disorders) | 47
Headache (Nervous system disorders) | 105
Insomnia (Psychiatric disorders) | 54
Proteinuria (Renal and urinary disorders) | 102
Cough (Respiratory, thoracic and mediastinal disorders) | 57
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 131
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 153
Alopecia (Skin and subcutaneous tissue disorders) | 143
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 79
Hypertension (Vascular disorders) | 369

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2012-02-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT01571284/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT01571284/SAP_001.pdf